CLINICAL TRIAL: NCT03057210
Title: Effects of Massage on the Short-term Post-exercise Recovery on Functional, Clinical and Metabolic Outcomes
Brief Title: Effects of Massage on the Short-term Post-exercise Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SaoPSU3
Record Dates: First submitted 2017-01-30; First posted 2017-02-20 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers
Keywords: Exercise; Massage; Post-exercise recovery; Athletic performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- S1 (Basal) (No Intervention): The behavior of the variables of functional and clinical outcome will be analyzed under no stress or recovery technique. In this stage, only the functional tests and the collection of clinical data will be performed.
- S2 (Massage) (Experimental): The behavior of the variables of functional and clinical outcome will be analyzed under stress or recovery technique. In this stage, only the functional tests and the collection of clinical data will be performed.
  Interventions: Other: Massage Protocol
- S3 (Exercise) (Experimental): The behavior of the variables of functional, clinical and metabolic outcome will be analyzed before the exercise protocol is performed. In this stage the volunteers will first perform the protocol for exhaustion, and in specific moments the blood lactate and clinical data will be collected, and 2h after the beginning of the exercise protocol, the functional tests will be performed.
  Interventions: Other: Stress Protocol
- S4 (Exercise + Immediate Massage) (Experimental): In this stage, the behavior of the variables of functional, clinical and metabolic outcome will be analyzed from the exercise protocol, followed by massage. Firstly the volunteers will carry out the protocol for exhaustion and the massage application will be done immediately after the end of the exercise. Blood lactate and clinical data will be collected at specific times during this stage. After 2h of the beginning of the stress protocol, the functional tests will be performed.
  Interventions: Other: Stress Protocol; Other: Massage Protocol
- • S5 (Exercise + Active Recovery + Delayed Massage) (Experimental): In this stage, the behavior of the variables of functional, clinical and metabolic outcome will be analyzed before the exhaustion protocol and the application of the massage after 1h of passive recovery. Firstly the volunteers will perform the protocol for exercise, followed by a passive recovery of 1h and then the massage application. The functional tests will be performed 2 hours after the stress protocol begins. Again, blood lactate collection and clinical data will occur at specific times.
  Interventions: Other: Stress Protocol; Other: Massage Protocol

INTERVENTIONS:
Other: Stress Protocol — Participants will be submitted to an exercise protocol consisting of a jumping program and a maximum short cycle test (ALMEIDAetal). The jumping program consists of 10 sets of 10 jumps with one minute interval between sets. The participants will then perform the Wingate Anaerobic Test protocol, which will be performed on a Biotec 2100 cycle ergometer (Cefise, Nova Odessa, Brazil). A 5-minute warm-up will be carried out where the participant will pedal at a speed of 60 to 90 rpm with a fixed load of 1.0 kg and perform sprints in the 2nd and 4th minute and the test itself, which consists of a maximum of pedals In 30 seconds with a stipulated load of 0.075 kP · kg-1 of the participant's body mass.
  Arms: S3 (Exercise); S4 (Exercise + Immediate Massage); • S5 (Exercise + Active Recovery + Delayed Massage)
Other: Massage Protocol — the present protocol will have a total of 12 minutes duration, being six minutes in the anterior region of the thigh (three minutes for each limb) and six minutes in the posterior region of the trunk.
  Surface and deep sliding techniques will be used, the latter being presented in two intensities, moderate or intense, gradually increased. The massage will be performed towards the muscle fibers, from distal to proximal and following the lymphatic flow. In addition to the standardization of the intensity of the massage performed by the physiotherapist, in order to avoid causing discomfort and possible variations in the application of the technique, participants should report their level of comfort from a scale that considers the technique "light", "moderate" or "Intense", corresponding respectively to surface slip, Deep Slip 1 and Deep Slip 2.
  Arms: S2 (Massage); S4 (Exercise + Immediate Massage); • S5 (Exercise + Active Recovery + Delayed Massage)

SUMMARY:
Objectives: To analyze the behavior of the effects of massage on clinical, metabolic and functional variables in different scenarios: i) under no stress or massage application; ii) after massage; iii) after exhaustion protocol; iv) after the immediate application of post-exercise massage; v) after application of the massage 1hour post-exercise.

Method: This was a randomized cross-over clinical trial in which 24 participants had their clinical, functional and metabolic outcome data analyzed under different scenarios: i) control scenario (CO): basal condition (under no stress or massage application); ii) Massage (MA): after receiving the massage; iii) Exhaustion protocol (PE): after protocol of exhaustion; iv) PE + immediate massage (EMI): after the protocol of exhaustion followed immediately by massage; iv) PE + delayed massage (EMT): after the protocol of exhaustion and massage received 1h after its end. The exhaustion protocol used consisted of 10 series of 10 jumps and one Wingate test and the manual massage protocol was composed of 12 minutes of massage, 3 minutes for the anterior region of the thigh of each lower limb and 6 minutes to the dorsal trunk. The variables studied were: muscle soreness, perceived recovery, maximal voluntary isometric contraction (MVIC), strength and power in the guided bar, vertical jump and blood lactate concentration [Lac].

Measurements. The primary outcome measures will be measured 2h after the start of each stage, and the secondary outcome measures will be measured at specific times during each stage. The primary outcome includes measures of functional performance, and the measures of secondary outcome includes clinical and metabolic variables.

DETAILED DESCRIPTION:
Introduction: Background: Massage has been shown over the years a recuperative technique widely used in sports. Studies demonstrate divergent results of the technique in terms of recovery of functional, clinical and metabolic performance after exercise. The wide methodological variety of these studies, as in relation to the moment of massage application, may be a possible justification for such a scenario. Thus, the study investigating the effects of massage applied at different moments of post-exercise recovery deserves to be highlighted.

Objectives: To analyze the behavior of the effects of massage on clinical, metabolic and functional variables in different scenarios: i) under no stress or massage application; ii) after massage; iii) after exhaustion protocol; iv) after the immediate application of post-exercise massage; v) after application of the massage 1hour post-exercise.

Design: A cross-over randomized clinical trial.

Method: This was a randomized cross-over clinical trial in which 24 participants had their clinical, functional and metabolic outcome data analyzed under different scenarios: i) control scenario (CO): basal condition (under no stress or massage application); ii) Massage (MA): after receiving the massage; iii) Exhaustion protocol (PE): after protocol of exhaustion; iv) PE + immediate massage (EMI): after the protocol of exhaustion followed immediately by massage; iv) PE + delayed massage (EMT): after the protocol of exhaustion and massage received 1h after its end. Exhaustion protocol: consisted of 10 series of 10 jumps and one Wingate test. Manual massage protocol: was composed of 12 minutes of massage, 3 minutes for the anterior region of the thigh of each lower limb and 6 minutes to the dorsal trunk.

Measurements. The primary outcome measures will be measured 2h after the start of each stage, and the secondary outcome measures will be measured at specific times during each stage. The primary measures includes the Strength and power test, Maximal voluntary isometric contraction (MVIC) and Squat jump. The secondary measures includes the subjective pain assessment, perception of recovery, psychological questionnaire, belief questionnaire and de analysis blood lactate concentration.

The variables studied were: muscle soreness, perceived recovery, maximal voluntary isometric contraction (MVIC), strength and power in the guided bar, vertical jump and blood lactate concentration [Lac].

Analysis: The normality of the data will be evaluated through the Shapiro-Wilk test. The sphericity of the data was tested by the Mauchly's test. In case of breach of the sphericity assumption, Greenhouse-Geisser corrections were used. Effect size was calculated using partial eta-square (η²) and interpreted as small (≥0.01), moderate (≥0.06) or large (≥0.14). When identified a large effect size, was used the Friedman's test with post-hoc Bonferroni test, for soreness and perceived recovery, and Repeated Measures ANOVA with post-hoc Tukey's test for vertical jump and MVIC. The level of significance was set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (self-report)
* Male gender;
* Aged between 18-30 years;

Exclusion Criteria:

* Presence of anemia, inflammation, or diabetes;
* History of muscle injury in the lower limbs or trunk in the previous six months;

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Squat jump | In Stage 1 (Baseline), 2 hours after the intervention in Stage 2, and 2 hours after the stress protocol in Stages 3, 4 and 5.
  For the initial positioning of the test, the participant was instructed to remain with the soles of the feet in contact with the jump platform (Multisprint, Hidrofit, Brazil), lower limbs flexed at 90º, hands at waist, trunk erect and without previous movements. Participants were familiarized with the test procedures, and were instructed to perform a maximum jump keeping the knees extended (180º of angulation)(27). Each participant performed three jumps with rest interval of 30 seconds between them and the best measure was adopted.
Maximal voluntary isometric contraction (MVIC) | In Stage 1 (Baseline), 2 hours after the intervention in Stage 2, and 2 hours after the stress protocol in Stages 3, 4 and 5.
  Prior to the MVIC assessment, the participants performed a warm-up consisting of 10 repetitions of knee flexion-extension at 180°.s-1 (3.14rad.s-1) throughout all the range of motion(28). Muscle function was determined by the highest torque normalized by participants' body weight (MVIC/weight), obtained through MVIC of the knee extensors of the dominant limb positioned at 60º of knee flexion (with 0º corresponding to the maximum extension) in the isokinetic dynamometer (Biodex System 4 Pro, New York, USA). Participants were instructed and verbally encouraged to perform maximal contractions during the test. There were 2 minutes of rest between the repetitions.
Strength test | In Stage 1 (Baseline), 2 hours after the intervention in Stage 2, and 2 hours after the stress protocol in Stages 3, 4 and 5.
  In a vertical squat with a guided bar, the participants performed squats with continuous movement until the thighs reached the horizontal plane, with the trunk as aligned as possible, and immediately performed the opposite movement, returning to the initial position. For the strength test, the heating was composed of 10 repetitions at 40% of the body mass of the participants. The last trunk extension performed without compensations with the highest possible load was determined as 1RM (one-repetition maximum). There were 2 minutes of rest between sets.
Power test | In Stage 1 (Baseline), 2 hours after the intervention in Stage 2, and 2 hours after the stress protocol in Stages 3, 4 and 5.
  In a vertical squat with a guided bar, the participants performed squats with continuous movement until the thighs reached the horizontal plane, with the trunk as aligned as possible, and immediately performed the opposite movement, returning to the initial position. The distance performed eccentrically and the concentric velocity of each repetition were recorded by a linear velocity transducer. The eccentric phase was performed at a controlled mean velocity of 0.5 m/s and the concentric phase at maximum velocity (explosively). The warm up was composed of five repetitions with the bar (14 kg) and the test was performed progressively and with increments of 10 kg in each series, with two attempts performed with each load until the participant reached the load closest to his 1RM. There was a 2-minute interval between repetitions. The best attempt with each load was recorded.

SECONDARY OUTCOMES:
Psychological questionnaire | In stages 1 to 5 at the beginning of the session before the interventions
  Participants were invited to fill out a psychological questionnaire that aims to subjectively document physical and mental readiness scores for exercise, fatigue, vigor, drowsiness, and muscle pain. It is important to inform that the intention of the application of this instrument was to provide control data on the general condition of the volunteer at the beginning of each session and not the verification of effects related to the interventions proposed in this trial.
  Thus, participants were instructed to mark a dash on a 10-centimeter visual analog scale between two extremes, zero being "least possible" and 10 indicating "most possible" for each rating.
Belief Questionnaire | In stages 1 to 5 at the beginning of the session before the interventions
  Participants were invited to respond to a questionnaire designed to measure beliefs about the effectiveness of the technique they were exposed to. It is an adaptation of the questionnaire used in the study by Moraska et al. (20). In this questionnaire participants were instructed to respond with "Yes", "No" or "I do not know" the following question: "Do you think massage will be beneficial to your recovery after intense exercise?"
Blood lactate concentration - [Lac] | Baseline and at minutes 2, 5, 8, 11, 14, 30, 60, 90 and 120 after the stress protocol in stages 3, 4 and 5.
  For analysis of blood lactate concentration [Lac], 25 μl of the ear lobe arterialized blood were collected from heparinized capillaries and scrounged in eppendorf-type polyethylene tubes (1.5 mL) containing 50 μl of sodium fluoride (NaF - 1%), for later lactacidemic analysis, performed in a laximeter (YSI, Yellow Springs - 1500, OH, USA). The lactate values were expressed in mmol / L. The lactate curve was analyzed from the absolute plasma lactate values. Blood lactate samples were collected prior to the initiation of the exhaust protocol, and at minutes 2, 5, 8, 11, 14, 30, 60, 90 and 120 after the protocol of physical exhaustion, and therefore comprising at some moments the period of performing the massage.
Subjective pain assessment | In Stages 3, 4 and 5: in the minutes 13, 60, 73 and 120 after the stress protocol.
  The subjective evaluation of pain was obtained through the Visual Analogue Scale (VAS), graded from 0 to 10, with zero being the total absence of pain and 10 the maximum level of pain supported by the individual. The participants were asked to perform an isometric contraction of the dominant quadriceps muscle, and the subjects were asked about the presence of pain in this limb, identifying by means of the scale the number corresponding to the intensity of pain at the present moment.
Perceived recovery | In Stages 3, 4 and 5: in the minutes 13, 60, 73 and 120 after the stress protocol.
  Perceived recovery of lower limbs submitted to PEF was assessed by a 10-point Likert Scale, where 1 indicates "not recovered" and 10 "fully recovered".
  The scale was presented to the participants and so that they were not influenced by the researcher, they answered the following question: "From 1 to 10 points, how do you rate your perception of recovery felt in your lower limbs if you had to do the same exercise protocol at this time? "

CONTACTS AND LOCATIONS:
Locations (1):
- Malu Dos Santos Siqueira, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No